CLINICAL TRIAL: NCT06565780
Title: Evaluation of the Performance and Safety of the Aktiia Spot-check Optical Blood Pressure Monitoring (OBPM) Device At Wrist Against Double Auscultation: a Multicentric Prospective Clinical Study
Brief Title: Evaluation of the Performance and Safety of the Aktiia Spot-check Optical Blood Pressure Monitoring Device At Wrist Against Double Auscultation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aktiia SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OBPM_FOX2024
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Aktiia.product-G0 device under test (Other): Subjects will be asked to stay seated while blood pressure and pulse rate measurements are taken at different timepoints with the device under test and references.
  Interventions: Device: Device under test evaluation against references

INTERVENTIONS:
Device: Device under test evaluation against references — Subjects will be asked to stay seated while blood pressure and pulse rate measurements are taken at different timepoints with the device under test and references.
  Device under Test: Aktiia.product-G0 References: Cuff for double auscultation for blood pressure and Electrocardiogram for pulse rate.

SUMMARY:
This study, with N = 85 participants minimum over 3 visits spread over 23 hours, has been designed to assess the accuracy and precision of the Blood Pressure and pulse rate values as generated by Aktiia.product-G0 for up to 23 hours after initialization in a cohort of subjects representative of the US population.

For the study, subjects will be asked to stay seated while measurements are taken at different timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide an informed consent to participate.
2. Participant must be willing and able to comply with all of the study procedures and return for a day 2 visit.
3. Participants must be 22 to 59 years of age.
4. Participant or witness must be able to read or write in English.

Exclusion Criteria:

1. Participants with compromised circulation, injury, or physical malformation of the equipment test sites or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the sites utilized.)
2. Female participants who are known to be pregnant or who are trying to get pregnant confirmed by a day 1 positive urine pregnancy test unless the study participant is known to be not of child-bearing potential.
3. Participants with known clotting disorders or currently taking a prescription blood thinner.
4. Other known health conditions that will prevent safe participation in the study upon disclosure in Health Assessment Short Form or verbally.
5. Participants suffering from sustained cardiac arrhythmias that can lead to weak or unstable pressure pulses including tachycardia (heart rate at rest > 120bpm) and atrial fibrillation.
6. Participants suffering from pathologies that systematically reduce peripheral perfusion including Raynaud's disease, diabetes, renal dysfunctions (eGFR < 60mL / min / 1.73 m2), hyper- / hypothyroidism, pheochromocytoma or arteriovenous fistula.
7. A wrist circumference below 14 cm or above 23 cm.
8. An upper arm circumference < 22cm or > 42cm.
9. Any subject that, in the opinion of the investigator, does not exhibit any phenotype relevant to the objectives of this study.
10. Any condition or circumstance that, in the opinion of the investigator, may preclude study completion, interfere with accurate data collection, bias the results, by instance a subject presenting a lateral Blood Pressure difference at screening of more than 15 mmHg for the systolic and/or more than 10 mmHg for the diastolic.

Ages: 22 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Blood pressure mean value of differences | 23 hours
  The mean value of the differences between Aktiia.product-G0 and double auscultation blood pressure measurements.
Blood pressure standard deviation of differences | 23 hours
  The standard deviation of the differences between Aktiia.product-G0 and double auscultation blood pressure measurements.

SECONDARY OUTCOMES:
Heart rate root-mean-square error | 23 hours
  The root-mean-square difference between the Aktiia.product-G0 heart rate determinations and the reference method.

CONTACTS AND LOCATIONS:
Locations (1):
- Parameters Research Laboratory, Broomfield, Colorado, United States